CLINICAL TRIAL: NCT04845022
Title: Incidence of Snakebite Associated Thrombotic Microangiopathy & Role of Peripheral Blood Smear as a Predictor of Clinical Outcome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jubilee Mission Medical College and Research Institute (Other)
Responsible Party: Principal Investigator, MAGLIN TOMY, Junior Resident, Jubilee Mission Medical College and Research Institute
Other Study IDs: 16/21/IEC/JMMC&RI
Record Dates: First submitted 2021-04-10; First posted 2021-04-14 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: SNAKEBITE; THROMBOTIC MICROANGIOPATHY; SCHISTOCYTES
Keywords: TMA, Peripheral blood smear(PBS)
MeSH Terms: conditions — Snake Bites; Thrombotic Microangiopathies; Sickle Cell Trait

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to find the overall incidence of thrombotic microangiopathy in snakebite victims. As we know snakebite is a common in tropical regions. Many a times the early diagnosis of TMA is missed and precious time which could have helped in improving the patient prognosis is lost. Also via this study we wish to learn the role of cost effective test like peripheral smear which could help learn morphological picture of red blood cells and thus help in early prediction of patients clinical prognosis.

DETAILED DESCRIPTION:
All snakebite patients brought to emergency department with history of bite and prolonged whole blood clotting time (WBCT) will be included in the study . their samples for hemogram, RFT and LDH would be collected in corresponding tubes . from sample for hemogram a peripheral blood smear (PBS) would be prepared , also the sample would be checked for direct coomb's test (DCT) positivity. DCT positive patients would be excluded from study . Also patients who received blood or blood components from outside hospital or patients with known history of hemolytic disease or patients on anti platelets or anticoagulants would also be excluded from this study .

thus patients who meet the exclusion and inclusion criteria would be followed up after 48 hours and their hemogram , RFT and LDH would be re assessed to check for presence of hemolysis , thrombocytopenia and acute kidney injury(AKI) .From the hemogram sample PBS would be prepared to check for presence of schistocytes.

Here we aim to study for incidence of TMA - defined as presence of MAHA( microangiopathic hemolytic anemia ) , thrombocytopenia and presence of AKI . MAHA is detected as drop of hb, presence of schistocytes in PBS , increase in LDH and increase in retic count. India is a tropical country and the southern state of Kerala , this study is done with the purpose of finding the prevalence of TMA among patients of snakebite brought to a tertiary care centre. Most often the victims are farmers or people from middle class. A cost effective test such as peripheral smear can help in predicting the prognosis and thereby aid in deciding whether the patient should require a multi disciplinary treatment early on and thereby play a pivotal role in saving patient life as well as provide an economical solution.

ELIGIBILITY:
Inclusion Criteria:

* All patients with a history of snakebite and with prolonged WBCT.

Exclusion Criteria:

* Patients administered with blood or blood components prior to admission
* Known case of bleeding disorders
* Known case of haemolytic anaemia
* Patients on antiplatelets or anticoagulants

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All snakebite victims who meet the inclusion criteria would be included in the study
Sampling Method: Probability Sample
Enrollment: 81 (Estimated)
Dates: Start 2021-01-28 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
To find the number of peripheral smear samples of TMA snakebite in which schistocyte grading helps in predicting the patient clinical outcome | 1 year
  To find the number of PBS smears in which morphological evaluation of RBC in PBS examination helps in predicting clinical outcome in snakebite associated TMA

SECONDARY OUTCOMES:
To find the number of hematotoxic snakebites associated with thrombotic microangiopathy (TMA) cases within 7days of admission | 1 year
  To find the number of TMA amongst snakebite victims in population coming to a tertiary care center in Kerala

CONTACTS AND LOCATIONS:
Overall Officials: Aboobacker Rafi, MD, Study Chair — Jubilee Mission Medical College and Research Institute
Locations (1):
- Jubilee Mission Medical College, Thrissur, Kerala, India